CLINICAL TRIAL: NCT04594161
Title: Effectiveness of Drainage of the Kidney by Percutaneous Nephrostomy Catheter Placement Vs. Retrograde Double J Catheter Placement in Patients With Symptoms of Obstructive Kidney Disease Caused by Urolithiasis
Brief Title: Effectiveness of Drainage by PCN vs. JJ in Patients With Symptoms of Obstructive Kidney Disease Caused by Urolithiasis
Acronym: STONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Alrijne Hospital (Other)
Responsible Party: Principal Investigator, Prof.dr. H.P. Beerlage, Professor doctor H.P. Beerlage, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: METC 2020_057; NL70822.058.19 (Other: ABR)
Record Dates: First submitted 2020-07-16; First posted 2020-10-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Urolithiasis; Urologic Diseases; Urinary Calculi; Urinary Obstruction; Urinary Stone; Ureteric Obstruction; Calculus Ureteral; Stone Ureter; Stone;Renal; Stone, Kidney; Stone, Urinary; Obstruction Ureter; Obstruction; Ureter Calculi; Ureter Obstruction; Kidney Diseases; Kidney Calculi; Kidney Failure, Acute; Kidney Dysfunction; Kidney Insufficiency; Pyelonephritis; Pyelonephritis Acute; Pyelonephritis Obstructive; Pyelonephritis; Calculus; Pyelonephritis; Obstruction; Pyelonephrosis; Hydronephrosis; Hydronephrosis; Infection; Hydronephrosis, Infected; Hydronephrosis; Obstruction, Ureter; Hydronephrosis; Obstruction, Renal Calculus; Hydronephrosis, Secondary; Renal Pelvis; Obstruction
Keywords: Urolithiasis; Urologic Diseases; Urinary Calculi; Urinary Obstruction; Urinary Stone; Nephrostomy; Complications; Catheter Complications; double j catheter; JJ catheter; urinary stent; percutaneous nephrostomy; stent
MeSH Terms: conditions — Urolithiasis; Urologic Diseases; Urinary Calculi; Ureteral Obstruction; Ureterolithiasis; Nephrolithiasis; Kidney Calculi; Bites and Stings; Kidney Diseases; Acute Kidney Injury; Renal Insufficiency; Pyelonephritis; Calculi; Hydronephrosis; Infections; Pyonephrosis; Neoplasm Metastasis | interventions — Nephrostomy, Percutaneous; Nephrotomy; Stents

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Masking Description: No masking is possible because stent is visible to patient and physician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Nephrostomy (Active Comparator): drainage of the kidney by means of a percutaneous Nephrostomy
  Interventions: Device: Percutaneous Nephrostomy
- Double J catheter (Active Comparator): drainage of the kidney by means of a double J catheter
  Interventions: Device: Double J catheter

INTERVENTIONS:
Device: Percutaneous Nephrostomy — A Percutaneous Nephrostomy will be placed in patients with obstructive urolithiasis
  Other Names: PCN; Nephrostomies, Percutaneous; Percutaneous Nephrostomies; Nephrostomy
  Arms: Percutaneous Nephrostomy
Device: Double J catheter — A Double J catheter will be placed in patients with obstructive urolithiasis
  Other Names: stent; JJ; internal stent; JJ catheter; urinary stent; internal urinary stent; ureteral stent; internal ureteral stent; internal ureteric stent; ureteric stent; ureteral stents; internal ureteral stents; internal ureteric stents; ureteric stents; double j ureteral catheter; double-j catheter; internalized double-j catheter
  Arms: Double J catheter

SUMMARY:
To investigate the effectiveness of percutaneous nephrostomy catheter placement versus retrograde double J catheter placement in patients with symptoms of obstructive kidney disease (with either infection and/or pain and/or kidney function deterioration) caused by urolithiasis.

DETAILED DESCRIPTION:
SUMMARY Rationale If a stone obstructs the ureter and impairs urine-efflux from the kidney this may cause infection, pain resulting from a renal colic and/or renal impairment. Drainage of the kidney may be necessary and can be established by placement of either a percutaneous nephrostomy (PCN) or a retrograde double J catheter (JJ). Considering method of drainage, setting, room in which drainage procedures takes place and anesthesia method, there are in fact 16 different approaches for drainage available, each with its own consequences for the patient and on expenses. Although evidence is poor, both methods of drainage are to be considered as equal.[1] This is reflected by the differences in preference between different countries.[2] In 2016 the Dutch association for urology (Nederlandse Vereniging voor Urologie (NVU)) marked this subject as one of the primary knowledge gaps in urology in The Netherlands and gave it priority on the national knowledge agenda for urology.[3] From patients' as well as from societal perspective it is of importance that the decision for placement of either PCN or JJ will be made based on evidence based arguments and in a uniform way.

Hypothesis: Percutaneous nephrostomy is non inferior to retrograde double J catheter regarding time to clinical recovery. Secondly, patient reported outcome measures (PROMS) comparing treatment room and OR settings of drainage procedures will most likely not be significantly different.

Finally, because percutaneous nephrostomy catheters are more often placed in a (outpatient) urological or radiological treatment room, this is expected to be less expensive than placement of a double J catheter (more often placed in the OR). Objective: To investigate the effectiveness of percutaneous nephrostomy catheter placement versus retrograde double J catheter placement in patients with symptoms of obstructive kidney disease (with either infection and/or pain and/or kidney function deterioration) caused by urolithiasis.

Study design: Multicenter prospective randomized controlled non-inferiority trial.

Study population: Male and female adult patients with signs of obstructive kidney disease with kidney or ureteral lithiasis as an underlying cause and with an indication for drainage based on symptoms of or laboratory tests indicating infection and/or pain and/or kidney function.

Intervention: One group receives drainage by percutaneous nephrostomy catheter placement as opposed to the other group which will receive drainage by retrograde double J catheter placement.

Main study parameters/endpoints:

The primary objective is to assess whether a PCN is non-inferior to double J catheter regarding time to clinical recovery in patients with obstructive kidney disease resulting from urolithiasis.

The primary outcome parameter is time to clinical recovery. Clinical recovery is defined as reaching one or more of the following criteria. The mandatory amount of criteria to achieve clinical recovery is dependent on the indication for placement of a PCN or a JJ.

* If indication for drainage is infection: improvement of infection, indicated by a decrease of WBC in two executive laboratory results and below 15.000 mm3 and a body temperature of 36-38.5 C. and/or
* If indication for drainage is untreatable pain: Numeric rating score (NRS) considering pain resulting from a renal colic is improved and < 3 points and/or
* If indication for drainage is deterioration of kidney function: improvement of creatinine/ Glomerular Filtration Rate (GFR) in two executive laboratory results It may occur that the indication for drainage is a combination of the above named indications. Clinical recovery will then be reached in case all parameters related to the different indications are within the set range. Secondary outcomes are further clinical data, PROMS (measured by the EQ-5D-5L, NRS, a satisfaction scale and a catheter questionnaire) and societal costs (measured by a diseasespecified iMCQ questionnaire).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The placement of either PCN or double J catheter is standard care. Currently the choice for PCN or a double J catheter is based on expert opinion and may be driven by arguments considering logistics or assumptions about the quality of life for a patient after placement.

Considering the difference in rate of placement of both PCN and double J catheter between various hospitals and different countries, it is believed experts have no uniform work method to handle the dilemma of choosing between these two techniques.[2] Furthermore the current EAU-guideline 2018 states that both methods of drainage are to be considered as equal.[1] Therefore there is no reason to believe, patients will be affected negatively by being placed randomly in either the double J group or the PCN group. Questionnaires will be filled in daily during hospitalization and twice or less afterwards. This is not considered to be a risk for the patient. The longest questionnaires (EQ-5D-5L and iMCQ) will take approximately 10-20 minutes to fill in, additional to the shorter scales (NRS, satisfaction scale) which will take approximately 1 minute to fill in. Generally It will take 90 minutes, spread over the course of three months, to fill in all questionnaires. For frequency and timing of the questionnaires. Finally, no additional visits to a hospital, withdrawal of blood samples or exposure to radiation is to be expected when taking part in this study.

ELIGIBILITY:
Inclusion Criteria:

- In order to be considered eligible to participate in this study, a subject must meet all of the following criteria:

* Male/female >18 year
* Symptoms and/or laboratory results indicating obstructive kidney disease with or without infection.
* A kidney or ureteral stone is present on ultrasound or CT (max 3 months old prior to presentation)
* Both drainage techniques are feasible and safe in opinion of the treating physician (from logistics point of view and in the best interest of the patient).
* Willing and able to comply with filling in questionnaires and follow-up regiment

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Analphabetic or not mastering the Dutch language
* Pregnancy
* Usage of anticoagulation agents other than acetylsalicylic acid.
* Contraindication for either technique looking at history and anatomy (e.g. kidney transplant, pouch, Bricker deviation, urethral or ureteral stenosis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
time (hours) to clinical recovery regarding infection | 3 months
  Unit is hours (0-∞), higher scores mean a worse outcome. Clinical recovery is defined as reaching one or more of the following criteria (all criteria are added seperately)
  - If indication for drainage is infection clinical recovery is defined as: improvement of infection, indicated by a decrease of WBC (unit: mm3) in two executive laboratory results and at least below 15.000 mm3.
time (hours) to clinical recovery regarding infection | 3 months
  Unit is hours (0-∞), higher scores mean a worse outcome. Clinical recovery is defined as reaching one or more of the following criteria (all criteria are added seperately)
  - If indication for drainage is infection clinical recovery is defined as: improvement of infection, indicated by a body temperatur between 36.0-38.5 °Celsius.
  and/or
  * If indication for drainage is untreatable pain: Numeric rating score (NRS) considering pain resulting from a renal colic is improved and < 3 points and/or
  * If indication for drainage is deterioration of kidney function: improvement of creatinine/ Glomerular Filtration Rate (GFR) in two executive laboratory results
time (hours) to clinical recovery regarding pain | 3 months
  Unit is hours (0-∞), higher scores mean a worse outcome. Clinical recovery is defined as reaching one or more of the following criteria (all criteria are added seperately) If indication for drainage is untreatable pain clinical recover is defined as: Numeric Rating Score (NRS) considering pain resulting from a renal colic is improved and < 3 points (higher scores mean greater level of pain).
time (in hours) to clinical recovery regarding kidney function | 3 months
  Unit is hours (0-∞), higher scores mean a worse outcome. Clinical recovery is defined as reaching one or more of the following criteria (all criteria are added seperately) If indication for drainage is deterioration of kidney function: improvement of creatinine (μmol/L) and/or Glomerular Filtration Rate (ml/min/1.73 m2) in two executive laboratory results.

SECONDARY OUTCOMES:
patient reported outcome measures (PROMS) quality of life | 3 months
  EQ-5D-5L questionnaire (range 0-1; greater scores reflect a higher quality of life).
patient reported outcome measures (PROMS) pain score | 3 months
  Numeric Rating Score (NRS) considering pain questionnaire (range 0-10; greater scores reflect higher pain levels)
patient reported outcome measures (PROMS) satisfaction | 3 months
  satisfaction scale (range 0-10; greater scores reflect higher levels of satisfaction)
patient reported outcome measures (PROMS) catheter related problems | 3 months
  catheter questionnaire. All answers will be analysed using frequencies. No score is applicable.
patient reported outcome measures (PROMS) cost and productivity | 3 months
  disease-specified iMCQ (Medical Consumption Questionnaire)/iPCQ (Productivity Cost Questionnaire). All answers will be analyzed using frequencies and will be used in economical models to calculate productivity burden and societal and individual costs.
patient reported outcome measures (PROMS) on costs iMCQ (Medical consumption questionnaire) | 3 months
  disease-specified iMCQ (Medical Consumption Questionnaire). All answers will be analyzed using frequencies and will be used in economical models to calculate productivity burden and societal and individual costs.
patient reported outcome measures (PROMS) productivity | 3 months
  iPCQ (Productivity Cost Questionnaire). All answers will be analyzed using frequencies and will be used in economical models to calculate productivity burden and societal and individual costs.

CONTACTS AND LOCATIONS:
Overall Officials: Ad Hendrikx, dr., Study Chair — no affiliation
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: official dutch website — https://zorgevaluatienederland.nl/stone